CLINICAL TRIAL: NCT02619539
Title: Shock Index To DEtect Low Plasma Fibrinogen In Trauma (SIDE)
Acronym: SIDE
Status: Completed | Type: Observational
Sponsor: Masaryk Hospital Krajská zdravotní a.s. (Other)
Responsible Party: Principal Investigator, Josef Skola, Dr., Masaryk Hospital Krajská zdravotní a.s.
Other Study IDs: KAPIM-1
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Trauma, Multiple
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma patients: All patients having / suspected to have severe trauma injuries admitted to participating centers.
  Interventions: Procedure: plasma fibrinogen measurement

INTERVENTIONS:
Procedure: plasma fibrinogen measurement — plasma fibrinogen measurement

SUMMARY:
Shock-index is potentially an easy tool to estimate the risk of hypofibrinogenemia without the need to perform other potentially time consuming investigations.

DETAILED DESCRIPTION:
Hypofibrinogenemia is common in severe trauma and below the threshold of 2.3 g/l is associated with increased mortality. Although guidelines for management of the trauma induced coagulopathy does not recommend any specific timing of fibrinogen substitution, several papers suggest that early substitution might be associated with improved outcome. Laboratory measurement of plasma fibrinogen level, thromboelastometry and/or its estimation based on base excess, hemoglobin level, Injury Severity Score or combinations require diagnostic procedures that are associated with with a certain time delay and prolongs the time to fibrinogen substitution.

ELIGIBILITY:
Inclusion Criteria:

* patient having / suspected to have severe trauma transported to participating centers by cooperating Emergency Medical System organizations

Exclusion Criteria:

* possible alterations of plasma fibrinogen level in the time of trauma (inflammatory disease, malignant disease, pregnancy)
* administration of fibrinogen containing products (fresh frozen plasma, fibrinogen concentrate, cryoprecipitate) before sampling blood for fibrinogen level
* circumstances possibly interfering with plasma fibrinogen level measurement (prior the administration of hydroxyethylstarches)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having / suspected to have severe trauma admitted to participating centres.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that have plasma fibrinogen <2.3 g.l-1 on admission among those with shock-index >1. | On admission

CONTACTS AND LOCATIONS:
Overall Officials: Josef Skola, Dr., Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (2):
- Czechia (2):
  - University Hospital in Plzen, Pilsen
  - Masaryk Hospital in Usti nad Labem, Ústí nad Labem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hagemo JS, Stanworth S, Juffermans NP, Brohi K, Cohen M, Johansson PI, Roislien J, Eken T, Naess PA, Gaarder C. Prevalence, predictors and outcome of hypofibrinogenaemia in trauma: a multicentre observational study. Crit Care. 2014 Mar 26;18(2):R52. doi: 10.1186/cc13798. PMID 24666991
- [Background] Spahn DR, Bouillon B, Cerny V, Coats TJ, Duranteau J, Fernandez-Mondejar E, Filipescu D, Hunt BJ, Komadina R, Nardi G, Neugebauer E, Ozier Y, Riddez L, Schultz A, Vincent JL, Rossaint R. Management of bleeding and coagulopathy following major trauma: an updated European guideline. Crit Care. 2013 Apr 19;17(2):R76. doi: 10.1186/cc12685. PMID 23601765
- [Background] Levy JH, Szlam F, Tanaka KA, Sniecienski RM. Fibrinogen and hemostasis: a primary hemostatic target for the management of acquired bleeding. Anesth Analg. 2012 Feb;114(2):261-74. doi: 10.1213/ANE.0b013e31822e1853. Epub 2011 Sep 29. PMID 21965371
- [Background] Schochl H, Maegele M, Solomon C, Gorlinger K, Voelckel W. Early and individualized goal-directed therapy for trauma-induced coagulopathy. Scand J Trauma Resusc Emerg Med. 2012 Feb 24;20:15. doi: 10.1186/1757-7241-20-15. PMID 22364525
- [Background] Schlimp CJ, Voelckel W, Inaba K, Maegele M, Ponschab M, Schochl H. Estimation of plasma fibrinogen levels based on hemoglobin, base excess and Injury Severity Score upon emergency room admission. Crit Care. 2013 Jul 12;17(4):R137. doi: 10.1186/cc12816. PMID 23849249